CLINICAL TRIAL: NCT00769223
Title: Pre-Operative Gleason Score and PSA and Clinical Stage in Predicting the Risk of Failure in Patients Undergoing Radiation Therapy for Localized Prostate Cancer
Brief Title: Predicting the Risk of Failure in Patients Undergoing Radiation Therapy for Localized Prostate Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CDR0000597000; H7056-08989 (Other: University of California, San Francisco); NCI-2019-08819 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 01558 (Other: University of California, San Francisco)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Radiation Toxicity
Keywords: radiation toxicity; recurrent prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage I prostate cancer; stage IV prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries | interventions — Brachytherapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Procedure: quality-of-life assessment
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Gathering information about the Gleason score, prostate-specific antigen (PSA) level, and cancer stage from patients who have undergone radiation therapy for prostate cancer may help doctors predict how patients respond to treatment and help plan the best treatment.

PURPOSE: This clinical trial is studying the Gleason score, PSA level, and cancer stage in predicting outcome in patients who have undergone radiation therapy for localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the value of the pre-operative Gleason score, prostate-specific antigen level, and clinical stage in predicting the risk of failure and death in patients who have undergone radiotherapy for localized prostate cancer.

OUTLINE: This is a multicenter study.

Patient medical records are reviewed to collect data about pre-treatment prostate biopsy, assigned Gleason score, prostate-specific antigen level, and radionucleotide bone scan.

Patients complete a Bowel Toxicity questionnaire to assess quality of life related to acute and long-term bowel toxicity after radiotherapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized adenocarcinoma of the prostate
* Has undergone radiotherapy (external beam radiotherapy and/or brachytherapy) with or without hormonal therapy for adenocarcinoma of the prostate in the University of California, San Francisco (UCSF) Radiation Oncology Department at San Francisco General Hospital or Veterans Administration Medical Center of San Francisco between 1987 and 2006

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate Cancer patients
Sampling Method: Probability Sample
Enrollment: 3561 (Actual)
Dates: Start 1993-02-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Value of the pre-operative Gleason score, prostate-specific antigen level, and clinical stage in predicting the risk of failure and death | Up to 30 years or until death
  The investigator will be analyzing the effect of baseline patient and clinical features such as age, Gleason score, PSA, clinical stage and percent positive biopsies on survival as well as quality of life parameters including potency, continence, and American Urological Association (AUA) symptoms scores

CONTACTS AND LOCATIONS:
Overall Officials: Mack Roach, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No